CLINICAL TRIAL: NCT03918889
Title: A Randomized Controlled Trial of the Effect of Dexmedetomidine Compared With Midazolam on Airway Reflex and Recovery Quality During Emergence From General Anesthesia After Partial and Total Laryngectomy
Brief Title: Effect of Dexmedetomidine in Preventing Cough and Postoperative Pain After Laryngeal Surgery for Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2013005
Record Dates: First submitted 2019-03-28; First posted 2019-04-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Laryngectomy; Status
Keywords: dexmedetomidine; midazolam; cough; sedation; pain
MeSH Terms: conditions — Cough; Pain | interventions — Dexmedetomidine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dexmedetomidine (Experimental): patients receive dexmedetomidine infusion
  Interventions: Drug: Dexmedetomidine Injectable Product
- midazolam (Experimental): patients receive midazolam infusion
  Interventions: Drug: Midazolam injection

INTERVENTIONS:
Drug: Dexmedetomidine Injectable Product — dexmedetomidine infusion at 0.5 µg•kg-1 for 10 min before tracheotomy then adjusted to 0.3µg•kg-1•h-1
  Arms: dexmedetomidine
Drug: Midazolam injection — midazolam infusion at 0.05 mg•kg-1 ten minutes before tracheotomy then adjusted to 0.02mg•kg-1•h-1
  Arms: midazolam

SUMMARY:
Background: During emergence from anesthesia for partial and total laryngectomy, severe airway reflex and systemic hypertension during recovery may lead to pneumoderm, hemorrhage, pneumomediastinum or pneumothorax. Dexmedetomidine is a selective α2-adrenoreceptor agonist that has sedative, analgesic, and sympatholytic properties. It has been reported dexmedetomidine can attenuate coughing reflex and prevent emergence agitation without delaying recovery and respiratory depression from general anesthesia. The purpose of this study was to investigate the effect of dexmedetomidine compared with midazolam on cough suppression and recovery quality during emergence from general anesthesia after partial and total laryngectomy.

Methods American Society of Anesthesiologists physical status I-II male adults undergoing elective laryngectomy under sevoflurane anesthesia were recruiting and randomly allocated to receive either dexmedetomidine(Group D, n = 60) infusion at 0.5 µg•kg-1 for 10 min before tracheotomy, then adjusted to 0.3µg•kg-1•h-1 or midazolam (Group M, n = 60) infusion at 0.05 mg•kg-1 ten minutes before tracheotomy, then adjusted to 0.02mg•kg-1•h-1. The primary outcome measure was the incidence and severity of cough. Hemodynamics, pain intensity [Visual Analogue Scale (VAS)] and Ramsay sedation scale (RSS) were also evaluated at awake, patients returning to ward from post anesthesia care unit (PACU),2h after surgery. postoperative sufentanil consumption, recovery time and the incidence of concerning adverse effects were recorded.

ELIGIBILITY:
Inclusion Criteria:

Subject scheduled for partial or total laryngectomy.

Exclusion Criteria:

Subject has respiratory disease; Subject has pharyngeal paraganglioma; Subject has cardiac disease; Uncontrolled hypertension; Subject has been taking β-adrenoreceptor blockers; Long-term abuse of alcohol (>6 months),opioids, or sedative-hypnotic drugs; Allergic to dexmedetomidine or midazolam; Subject has neuropsychiatric diseases; Operation time shorter than 1 h or longer than 4 h.

Ages: 35 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
The severity of cough | Time0:2hours after surgery
  Coughing severity was classified using the 3-point scale.:1=mild (single) cough, 2=moderate (≤5 s) cough, and 3=severe (>5 s) cough.

SECONDARY OUTCOMES:
HR | Time0: 0 minute after arriving the operation room
  Heart rate
SBP | Time0: 0 minute after arriving the operation room
  Systolic blood pressure
DBP | Time0: 0 minute after arriving the operation room
  Diastolic blood pressure
SpO2 | Time0: 0 minute after arriving the operation room
  Oxygen saturation using pulse oximetry
HR | Time1:0 minute after drug administration
  Heart rate
SBP | Time1:0 minute after drug administration
  Systolic blood pressure
DBP | Time1:0 minute after drug administration
  Diastolic blood pressure
SpO2 | Time1:0 minute after drug administration
  Oxygen saturation using pulse oximetry
HR | Time2:0 minute after intubation
  Heart rate
DBP | Time2:0 minute after intubation
  Diastolic blood pressure
SBP | Time2:0 minute after intubation
  Systolic blood pressure
SpO2 | Time2:0 minute after intubation
  Oxygen saturation using pulse oximetry
HR | Time3:0 minute after medicine intervention
  Heart rate
DBP | Time3:0 minute after medicine intervention
  Diastolic blood pressure
SBP | Time3:0 minute after medicine intervention
  Systolic blood pressure
SpO2 | Time3:0 minute after medicine intervention
  Oxygen saturation using pulse oximetry
HR | Time4:0 minute after laryngectomy
  Heart rate
DBP | Time4:0 minute after laryngectomy
  Diastolic blood pressure
SBP | Time4:0 minute after laryngectomy
  Systolic blood pressure
SpO2 | Time4:0 minute after laryngectomy
  Oxygen saturation using pulse oximetry
HR | Time5:0 minute after the completion of surgery
  Heart rate
SBP | Time5:0 minute after the completion of surgery
  Systolic blood pressure
DBP | Time5:0 minute after the completion of surgery
  Diastolic blood pressure
SpO2 | Time5:0 minute after the completion of surgery
  Oxygen saturation using pulse oximetry
HR | Time6:0 minute after awareness
  Heart rate
SBP | Time6:0 minute after awareness
  Systolic blood pressure
DBP | Time6:0 minute after awareness
  Diastolic blood pressure
SpO2 | Time6:0 minute after awareness
  Oxygen saturation using pulse oximetry
HR | Time7:0 minute after departure from the PACU
  Heart rate
SBP | Time7:0 minute after departure from the PACU
  Systolic blood pressure
BDP | Time7:0 minute after departure from the PACU
  Diastolic blood pressure
SpO2 | Time7:0 minute after departure from the PACU
  Oxygen saturation using pulse oximetry
Pain intensity | Time0:2hours after surgery
  Assessed by Visual Analogue Scale (VAS), (0, no pain; 10, the worst pain intolerable)
Sedation | Time0: 2hours after surgery
  Assessed by Ramsay sedation scale (RSS),1, Anxious or restless or both,2, Cooperative, orientated and tranquil,3,Responding to commands,4,Brisk response to stimulus,5,Sluggish response to stimulus,6, No response to stimulus.
the incidence of adverse effects | Time0:2hours after surgery
  desaturation,shivering,drowsiness, delirium,hypertension,hypotension,itching,arrhythmia,respiratory depression

CONTACTS AND LOCATIONS:
Overall Officials: Wenxian Li, PhD, Study Director — Department of Anesthesiology
Locations (1):
- Department of Anesthes iology, The Eye, Ear, Nose and Throat Hospital of Fudan University, Shanghai Medical College of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu R, Zhu Y, Lu Y, Li W, Jia J. Dexmedetomidine versus midazolam on cough and recovery quality after partial and total laryngectomy - a randomized controlled trial. BMC Anesthesiol. 2020 Sep 28;20(1):249. doi: 10.1186/s12871-020-01168-7. PMID 32988369